CLINICAL TRIAL: NCT00018369
Title: Mechanism of Aging-Related Changes in (HPA) Hydrocortisone Corticotropin Feedback Function
Brief Title: Age-Related Changes in Stress Hormone Regulation
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: AGCG-009-99F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Physiological Processes; Aging
Keywords: Aging; Hydrocortisone Corticotropin Feedback

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Studies investigating physiological processes involved in aging-related deficits in regulation of stress hormone systems.

ELIGIBILITY:
Exclusion Criteria:

* History of major psychiatric disorders,
* Neurologic disorder affecting cognitive function,
* Unstable medical problems,
* Medications including antidepressants, neuroleptics, anxiolytics, CNS stimulants, narcotic analgesics, anti-convulsants,
* Drugs effecting HPA axis function,
* Vision and hearing deficits,
* Undergoing major life event within one month or
* Loss of family member within 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dorin; Elaine Peskind; Alan Schatzberg; Joseph Belanoff
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States